CLINICAL TRIAL: NCT04466046
Title: The Effect on Anxiolytics With Type of Antiemetic Agents on Postoperative Nausea and Vomiting in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: The Effect on Anxiolytics With Type of Antiemetic Agents on Postoperative Nausea and Vomiting in High Risk Patients
Status: Completed | Type: Observational
Sponsor: Daegu Catholic University Medical Center (Other)
Responsible Party: Principal Investigator, Jung A, Assistant professor, Daegu Catholic University Medical Center
Other Study IDs: 19-100
Record Dates: First submitted 2020-07-02; First posted 2020-07-10 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PONV group: Patients with PONV after administration of midazolam 0.05mg/kg with ramosetron 0.3mg or palonosetron 0.075mg
- no PONV group: Patients with no PONV after administration of midazolam 0.05mg/kg with ramosetron 0.3mg or palonosetron 0.075mg

SUMMARY:
Nausea and vomiting after surgery are one of the complications that occur after general anesthesia, and the frequency is reported to range from 10% to 80% in the high-risk group. Several studies have introduced drugs and methods to prevent nausea and vomiting after surgery. Among them, midazolam administered before surgery is known to have anti-anxiolytic and sedative effects on the prevention of nausea and vomiting after surgery. It has also been reported to increase its effectiveness when administered with other antiemetic agents.

The purpose of this study is to compare the effects of administration of combination with midazolam and different antiemetic agents on the prevention of postoperative nausea and vomiting in high-risk patients.

DETAILED DESCRIPTION:
This prospective study evaluates female, nonsmoking patients undergoing laparoscopic cholecystectomy. The patients are divided into those with and without postoperative nausea and vomiting. The purpose of this study is to compare and observe the effect of administration of midazolam and two different antiemetics on prevention of postoperative nausea and vomiting.

0.05mg/kg of midazolam is administered intravenously 10 minutes before surgery as a pretreatment. 0.3mg ramosetron is administered intravenously right before the end of surgery and 0.075mg palonosetron is administered intravenously immediately after induction of anesthesia. The incidence of PONV, severity of nausea, use of rescue antiemetics, and pain severity was evaluated at 2 hours, 24hours, and 48 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* 20-65 years old with American Society of Anesthesiologists (ASA) physical status 1-2 and scheduled for laparoscopic cholecystectomy.

Exclusion Criteria:

* pregnant or breast feeding patients
* smokers
* patients with history of chronic opioid abuse
* hypersensitivity to 5-HT3 receptor antagonists or analgesics
* those who were antiemetic or opioid treatment within 24 hours prior to surgery

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: female patients aged 20 to 65 with ASA physical status 1 or 2 undergoing laparoscopic cholecystectomy
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
percentage of patients receiving ramosetron or palonosetron in each groups | 48 hours after surgery
  percentage of patients receiving ramosetron or palonosetron
severity of postoperative nausea in PONV group | 48 hours after surgery
  0 = none, 1 = mild, 2 = moderate, 3 = severe

SECONDARY OUTCOMES:
postoperative pain | 48 hours after surgery
  numerical analog scale : 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Jung A Lim, MD, Study Chair — Daegu Catholic University Medical Center
Locations (1):
- Daegu Catholic University Medical Center, Daegu, Nam-gu, South Korea

IPD SHARING:
Plan to Share IPD: No